CLINICAL TRIAL: NCT05526560
Title: A Prospective, Global Study Designed to Collect Real-world Clinical Outcomes of the MITRIS RESILIA Mitral Valve
Brief Title: Real-world Clinical Outcomes of the MITRIS RESILIA Mitral Valve
Acronym: MOMENTIS
Status: Active, not recruiting | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-09
Record Dates: First submitted 2022-08-25; First posted 2022-09-02 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Mitral Stenosis; Mitral Valve Insufficiency
Keywords: Mitral Valve Replacement
MeSH Terms: conditions — Mitral Valve Stenosis; Mitral Valve Insufficiency | interventions — Models, Biological

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients requiring replacement of their native or prosthetic mitral valve: Patients requiring replacement of their native or prosthetic mitral valve
  Interventions: Device: MITRIS RESILIA Mitral Valve, Model 11400M

INTERVENTIONS:
Device: MITRIS RESILIA Mitral Valve, Model 11400M — Replacement of mitral valve with MITRIS RESLIA Mitral Valve

SUMMARY:
Collect real-world data on acute and long-term safety and performance of the MITRIS RESILIA Mitral Valve, Model 11400M, in subjects requiring replacement of their native or prosthetic mitral valve with or without concomitant procedures.

DETAILED DESCRIPTION:
MOMENTIS is a prospective, observational, single-arm, multicenter global study designed to collect real-world clinical outcomes in up to 500 subjects who have received the MITRIS RESILIA Mitral Valve, Model 11400M.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at the time of informed consent
* Has a dysfunctional native or prosthetic mitral valve and requires mitral valve replacement surgery
* Provides written informed consent
* Willingness to follow protocol requirements

Exclusion Criteria:

* Active endocarditis 3 months prior to the procedure
* Stage 4 renal disease or requiring dialysis
* Less than 2-year life expectancy due to non-cardiovascular life-threatening disease
* High predicted risk of mortality prior to procedure

  * Society of Thoracic Surgeons (STS) Predicted Risk of Mortality (PROM) score of > 8 or
  * Surgeon estimated risk of mortality of > 8

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring replacement of their native or prosthetic mitral valve
Sampling Method: Non-Probability Sample
Enrollment: 504 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Freedom from valve related death or valve related reintervention | 1 year
  Freedom from valve related death or valve related reintervention at 1 year as determined by the Clinical Events Committee
Hemodynamic performance as measured by peak and mean gradient by echocardiography | 1 year
  Hemodynamic performance at 1 year as confirmed by echocardiography and Echo Core Lab evaluation

SECONDARY OUTCOMES:
Early rates of major cardiac events | 0 to 30 days
  Early (<=30 days) rates of major cardiac events
Late linearized rates of major cardiac events | >30 days and up through 10 years post implant
  Linearized rates of late (>30 days) major cardiac events
Functional improvement from baseline for New York Heart Association (NYHA) Class | Annually up to 10 years post implant
  Functional improvement from baseline for NYHA Class
Improvement from baseline for Quality of Life | 1, 3, 5, 8, and 10 years post implant
  Improvement from baseline for Quality of Life as measured by the Short Form (36) Health Survey (SF-36v2) (0-100 scale, with a higher score indicating less disability)

CONTACTS AND LOCATIONS:
Overall Officials: Gorav Ailawadi, MD, Principal Investigator — University of Michigan
Locations (34):
- United States (20):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Stanford University, Palo Alto, California
  - AdventHealth Orlando, Orlando, Florida
  - Piedmont Heart Institute, Athens, Georgia
  - Piedmont Heart Institute, Atlanta, Georgia
  - Ascension St. Vincent Heart Center, Carmel, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - Washington University Barnes-Jewish Hospital, St Louis, Missouri
  - Mount Sinai Hospital, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian Shadyside, Pittsburgh, Pennsylvania
  - Tristar Centennial Medical Center, Nashville, Tennessee
  - Ascension Saint Thomas, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Canada (4):
  - St. Paul's Hospital and Vancouver General Hospital, Vancouver, British Columbia
  - London Health Sciences Centre, University Hospital (LHSC), London, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec - Université Laval, Québec
- Germany (6):
  - Universitätsklinikum Augsburg, Augsburg
  - Rhoen-Klinikum Campus Bad Neustadt, Bad Neustadt an der Saale
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - University Clinic Bonn, Bonn
  - Klinikum Links der Weser, Bremen
  - Deutsches Herzzentrum München, München
- United Kingdom (4):
  - Royal Papworth Hospital, Cambridge
  - St. Thomas Hospital, London
  - King's College Hospital, London
  - Cleveland Clinic London, London

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers.